CLINICAL TRIAL: NCT02577133
Title: Prevention of Colic With the Probiotic Lactobacillus Reuteri in Mexican Infants: Randomized, Double-blind Study
Brief Title: Prevention of Colic With the Probiotic Lactobacillus Reuteri
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Principal Investigator, Dr. Jorge Ivan Valencia Moncada, Prevention of colic with the probiotic Lactobacillus reuteri DSM 17938 in Mexican infants: randomized, double-blind study, Hospital General Naval de Alta Especialidad - Escuela Medico Naval
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HGNAE-04
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Colic
Keywords: colic; probiotic; Lactobacillus reuteri; prevention
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus reuteri group (Active Comparator): Lactobacillus reuteri DSM 17938 1,000,000,000 CFU per day (5 drops) for 28 days
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938
- Placebo group (Placebo Comparator): Placebo (5 drops) for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — Lactobacillus reuteri DSM 17938 1,000,000,000 CFU per day (5 drops) for 28 days
  Other Names: BioGaia
  Arms: Lactobacillus reuteri group
Dietary Supplement: Placebo — The placebo consisted of an identical bottle with distilled water
  Arms: Placebo group

SUMMARY:
Colic is a term for inconsolable crying happened in the first months of life. Its etiology is multifactorial and caregiver and pediatrician generates among other problems: anxiety, risk of child abuse as well as economic costs.

There is now enough evidence for the treatment of colic using probiotics, especially Lactobacillus reuteri.

The investigators study aims to demonstrate the utility for the prevention of colic with L. reuteri and thereby avoid the problems caused by this pathology.

Objective: Compare the number of events of colic among infants with oral probiotic Lactobacillus reuteri during the first month of life versus infants with placebo

Study Design. Double blind, randomized, controlled, 492 neonates of 37-42 gestational age, breast or formula fed, will receive L. reuteri 5 drops (1x108 CFU) daily or placebo for 28 days. The investigators trial will be performed at Naval Hospital in Mexico City.

DETAILED DESCRIPTION:
Methods:

This study is planned for October 2015 to October 2016 aiming newborns born population in Naval Hospital

Inclusion:

* Term Healthy Newborns (RN) ≥38 weeks and ≤ 41 weeks of gestation
* Appropriate weight for gestational age
* ≥than 8 Apgar at 5 minutes
* Egress at the first 24-48 hours of life of the newborn with the mother of hospital
* No congenital or physical abnormalities on physical examination at birth.
* Availability during the study period.
* Thorough understanding of the protocol by parents
* Informed Consent is signed by both parents.

Exclusion:

* Administration of antibiotics to the mother for a week before the birth of the newborn.
* Administration of probiotics newborn before inclusion or consumption by the mother during these last two trimesters.
* Medication Management newborn different routine prescribed at birth.

Elimination

* Loss of monitoring
* Abandonment by parents
* Diagnosis of allergy to cow's milk protein (confirmed by resolution of symptoms after switching to Formula hypo allergenic or free feeding cow's milk by the mother in breastfed children).
* Diagnosis of structural alterations or gastrointestinal illness to explain the symptoms of colic in the following months after the inclusion

Interventions:

The patients enrolled will receive probiotics (1000000000 CFU per day) or placebo every days for 28 days

Weekly, each patient will be called twice to interrogate the number of events colic as well as the different variables under study

After birth, on 15, 30, 45 and 60 of life will be cited for clinical examination and review and weight dropper bottle of probiotic

• Principal: Number of events or inconsolable crying

• Secondary: Average or evacuations / day Average or regurgitation / day Drugs to decrease excessive crying Medical reviews for excessive crying Changes feeding for excessive crying Level of satisfaction with the care of the newborn (numerical scale from 0: the worst possible, 10: completely satisfied)

• Universal variables

Weight:

Size:

Gender Weeks gestation Type of birth Feeding of formula / breast-

ELIGIBILITY:
Inclusion Criteria:

* Term Healthy Newborns (RN) ≥38 weeks and ≤ 41 weeks of gestation.
* Appropriate weight for gestational age
* ≥than 8 Apgar at 5 minutes
* Egress at the first 24-48 hours of life of the newborn with the mother of hospital
* No congenital or physical abnormalities on physical examination at birth.
* Availability during the study period.
* Thorough understanding of the protocol by parents
* Informed Consent is signed by both parents.

Exclusion Criteria:

* Administration of antibiotics to the mother for a week before the birth of the newborn.
* Administration of probiotics newborn before inclusion or consumption by the mother during these last two trimesters.
* Medication Management newborn different routine prescribed at birth.

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 478 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Event number of colic | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Héctor Javier Varona Bobadilla, Dr., Principal Investigator — Secretaria de Marina-Armada de México (Mexican Navy)

REFERENCES:
- [Background] Hyman PE, Milla PJ, Benninga MA, Davidson GP, Fleisher DF, Taminiau J. Childhood functional gastrointestinal disorders: neonate/toddler. Gastroenterology. 2006 Apr;130(5):1519-26. doi: 10.1053/j.gastro.2005.11.065. PMID 16678565
- [Background] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956
- [Background] Douglas P, Hill P. Managing infants who cry excessively in the first few months of life. BMJ. 2011 Dec 15;343:d7772. doi: 10.1136/bmj.d7772. No abstract available. PMID 22174332
- [Background] E. Ortega Páeza , D. Barroso Espaderob Flashes pediátricos AEpap Cólico del lactante Rev Pediatr Aten Primaria Supl. 2013;(22):81-7
- [Background] Wolke D, Samara M, Alvarez Wolke M. Meta-analysis of fuss/cry durations and colic prevalence across countries: Proceedings of the11th International Infant Cry Research Workshop, June, 2011, The Netherlands.
- [Background] Cohen GM, Albertini LW. Colic. Pediatr Rev. 2012 Jul;33(7):332-3; discussion 333. doi: 10.1542/pir.33-7-332. No abstract available. PMID 22753793
- [Background] Barr RG, Rotman A, Yaremko J, Leduc D, Francoeur TE. The crying of infants with colic: a controlled empirical description. Pediatrics. 1992 Jul;90(1 Pt 1):14-21. PMID 1614771
- [Background] Romanello S, Spiri D, Marcuzzi E, Zanin A, Boizeau P, Riviere S, Vizeneux A, Moretti R, Carbajal R, Mercier JC, Wood C, Zuccotti GV, Crichiutti G, Alberti C, Titomanlio L. Association between childhood migraine and history of infantile colic. JAMA. 2013 Apr 17;309(15):1607-12. doi: 10.1001/jama.2013.747. PMID 23592105
- [Background] Savino F, Cordisco L, Tarasco V, Calabrese R, Palumeri E, Matteuzzi D. Molecular identification of coliform bacteria from colicky breastfed infants. Acta Paediatr. 2009 Oct;98(10):1582-8. doi: 10.1111/j.1651-2227.2009.01419.x. Epub 2009 Jul 9. PMID 19604166
- [Background] de Weerth C, Fuentes S, Puylaert P, de Vos WM. Intestinal microbiota of infants with colic: development and specific signatures. Pediatrics. 2013 Feb;131(2):e550-8. doi: 10.1542/peds.2012-1449. Epub 2013 Jan 14. PMID 23319531
- [Background] Savino F, Cresi F, Pautasso S, Palumeri E, Tullio V, Roana J, Silvestro L, Oggero R. Intestinal microflora in breastfed colicky and non-colicky infants. Acta Paediatr. 2004 Jun;93(6):825-9. PMID 15244234
- [Background] Iacono G, Merolla R, D'Amico D, Bonci E, Cavataio F, Di Prima L, Scalici C, Indinnimeo L, Averna MR, Carroccio A; Paediatric Study Group on Gastrointestinal Symptoms in Infancy. Gastrointestinal symptoms in infancy: a population-based prospective study. Dig Liver Dis. 2005 Jun;37(6):432-8. doi: 10.1016/j.dld.2005.01.009. Epub 2005 Mar 2. PMID 15893282
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Charrois TL, Sandhu G, Vohra S. Probiotics. Pediatr Rev. 2006 Apr;27(4):137-9. doi: 10.1542/pir.27-4-137. No abstract available. PMID 16581954
- [Background] http://www.biogaia.com/lactobacillus-reuter
- [Background] Talarico TL, Casas IA, Chung TC, Dobrogosz WJ. Production and isolation of reuterin, a growth inhibitor produced by Lactobacillus reuteri. Antimicrob Agents Chemother. 1988 Dec;32(12):1854-8. doi: 10.1128/AAC.32.12.1854. PMID 3245697
- [Background] Morelli L, Capurso L. FAO/WHO guidelines on probiotics: 10 years later. J Clin Gastroenterol. 2012 Oct;46 Suppl:S1-2. doi: 10.1097/MCG.0b013e318269fdd5. No abstract available. PMID 22955349
- [Background] Lifschitz C. Probiotics: Implications for Paediatric Health, Nestlé Nutrition Institute, South Asia Workshop Proceedings Vol. 1, Issue 1, 2013
- [Background] Savino F, Pelle E, Palumeri E, Oggero R, Miniero R. Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics. 2007 Jan;119(1):e124-30. doi: 10.1542/peds.2006-1222. PMID 17200238
- [Background] Savino F, Cordisco L, Tarasco V, Palumeri E, Calabrese R, Oggero R, Roos S, Matteuzzi D. Lactobacillus reuteri DSM 17938 in infantile colic: a randomized, double-blind, placebo-controlled trial. Pediatrics. 2010 Sep;126(3):e526-33. doi: 10.1542/peds.2010-0433. Epub 2010 Aug 16. PMID 20713478
- [Background] Chumpitazi BP, Shulman RJ. Five probiotic drops a day to keep infantile colic away? JAMA Pediatr. 2014 Mar;168(3):204-5. doi: 10.1001/jamapediatrics.2013.5002. No abstract available. PMID 24424486
- [Background] Sung V, Collett S, de Gooyer T, Hiscock H, Tang M, Wake M. Probiotics to prevent or treat excessive infant crying: systematic review and meta-analysis. JAMA Pediatr. 2013 Dec;167(12):1150-7. doi: 10.1001/jamapediatrics.2013.2572. PMID 24100440
- [Background] Indrio F, Di Mauro A, Riezzo G, Civardi E, Intini C, Corvaglia L, Ballardini E, Bisceglia M, Cinquetti M, Brazzoduro E, Del Vecchio A, Tafuri S, Francavilla R. Prophylactic use of a probiotic in the prevention of colic, regurgitation, and functional constipation: a randomized clinical trial. JAMA Pediatr. 2014 Mar;168(3):228-33. doi: 10.1001/jamapediatrics.2013.4367. PMID 24424513